CLINICAL TRIAL: NCT02775019
Title: Impact of the Daily Consumption of L.Reuteri-containing Lozenges on Oral and General Health in Crew Members of a Naval Ship at Sea
Brief Title: Health Impact of L.Reuteri Consumption in Crew Members of a Naval Ship at Sea
Acronym: NAVLAC16
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: German Naval Medical Institute (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ulrich Schlagenhauf, chairman Dept. of Periodontology, Wuerzburg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 02-2016-NAVLAC
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactobacillus reuteri lonzenges (Active Comparator): 2x daily repeated intake of lozenges containing 10E9 CFU Lactobacillus reuteri each for 42 days
  Interventions: Dietary Supplement: Lactobacillus reuteri
- Placebo lozenges (Placebo Comparator): 2x daily repeated intake of lozenges being void of Lactobacillus reuteri for 42 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri — 2 x daily repeated consumption of a lozenge containing 10E9 CFU Lactobacillus reuteri for 42 days
  Arms: Lactobacillus reuteri lonzenges
Dietary Supplement: Placebo — 2 x daily repeated consumption of a lozenge being void of Lactobacillus reuteri for 42 days
  Arms: Placebo lozenges

SUMMARY:
This study is designed to evaluate the impact of the regular consumption of probiotic Lactobacillus reuteri-containing lozenges over a period of 42 days on parameters of oral and general health in crew members of a naval ship at sea.

DETAILED DESCRIPTION:
Probiotic strains of Lactobacillus reuteri have demonstrated a significant impact on the composition of the oral and intestinal microbiome as well as modulating the host response in several clinical trials and in vitro experiments.

This two-arm double blind placebo controlled clinical trial will evaluate the impact of the regular consumption of L.reuteri-containing lozenges over a period of 42 days on parameters of oral and general health in crew members of a naval ship at sea.

2 x 36 healthy study subjects will be recruited from the crew members of the ship.

At baseline and at the end of the study (day 42) the following parameters will be recorded at the Ramfjord teeth (teeth 16, 21, 24, 36, 41, 44):

Bleeding on Probing (BoP) as the primary outcome

Secondary outcomes will be Gingival Index (GI) Plaque Control Record (PCR) Pocket Probing Depth (PPD) Pooled oral and intestinal (stool) microbial samples will be taken at baseline and at the end of the study for the subsequent analysis of the

* composition of the oral microbiome
* composition of the intestinal microbiome by whole genome sequencing

Furthermore the frequency of short-term sick leave due to respiratory or intestinal diseases among the study participants during the observation period will be recorded.

ELIGIBILITY:
Inclusion Criteria:

Minimum of 12 natural teeth

Exclusion Criteria:

Regular intake of antiinflammatory drugs affecting periodontal health (e.g. NSAIDs) Manifestation of systemic disease affecting periodontal health (e.g. diabetes) Use of antiseptic oral mouthrinses Drug/alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Bleeding on Probing | 42 days
  Number of sites being positive for bleeding on probing on the Ramfjord teeth (teeth 16, 21, 24, 36, 41, 44) with 6 probing sites per tooth

SECONDARY OUTCOMES:
Gingival Index (GI) | 42 days
  Recording of the GI on the vestibular and oral aspects of the Ramfjord teeth (teeth 16, 21, 24, 36, 41, 44)
Plaque Control Record (PCR) | 42 days
  Recording of the PCR on the vestibular and oral aspects of the Ramfjord teeth (teeth 16, 21, 24, 36, 41, 44)
Probing Pocket Depth (PPD) | 42 days
  Recording of the PPD at the Ramfjord teeth (teeth 16, 21, 24, 36, 41, 44) with 6 probing sites per tooth
Composition of the oral microbiome | 42 days
  Collection of pooled bacterial biofilm samples from the Ramfjord teeth for subsequent analysis by whole genome sequencing
Composition of the intestinal microbiome | 42 days
  Collection of microbial stool samples for subsequent analysis by whole genome sequencing
Short-term sick leave | 42 days
  Recording of the incidence of short-term sick leave due to gastrointestinal or respiratory diseases

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schlagenhauf, Prof. Dr., Principal Investigator — Chairman Dept. of Periodontology, University Hospital Wuerzburg, Germany
Locations (1):
- German Naval Medical Institute, Kronshagen, Germany

IPD SHARING:
Plan to Share IPD: Undecided